CLINICAL TRIAL: NCT03925545
Title: VisiOn Restoration With the FluidVisION AIOL
Brief Title: VisiOn Restoration With FluidVisION Accommodating Intraocular Lens (AIOL)
Acronym: ORION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PowerVision (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Device Feasibility
Other Study IDs: CTP07700
Record Dates: First submitted 2019-04-15; First posted 2019-04-24 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Unilateral (Experimental): Implantation with the FluidVision AIOL in one eye during cataract surgery. Only one eye was treated.
  Interventions: Device: FluidVision AIOL; Procedure: Cataract surgery
- Contralateral (Experimental): Implantation with the FluidVision AIOL in the first eye during cataract surgery, followed by implantation with the AcrySof IQ monofocal IOL in the fellow eye during a subsequent cataract surgery
  Interventions: Device: FluidVision AIOL; Device: AcrySof IQ monofocal IOL; Procedure: Cataract surgery

INTERVENTIONS:
Device: FluidVision AIOL — Investigational implantable medical device intended for long-term use over the lifetime of the cataract subject
Device: AcrySof IQ monofocal IOL — Commercially available implantable medical device intended for long-term use over the lifetime of the cataract subject
  Arms: Contralateral
Procedure: Cataract surgery — Standard cataract extraction with phacoemulsification

SUMMARY:
The objective of this study is to obtain an initial assessment of the safety and performance of an investigational AIOL in patients undergoing cataract extraction and IOL implantation.

DETAILED DESCRIPTION:
This study was originally designed as a single arm, unilateral study (one eye, one product only) to obtain an initial assessment of the safety and performance of an investigational IOL in subjects undergoing cataract extraction and IOL implantation. The study design was later modified to a contralateral study (both eyes, different product in each eye) to compare the safety and performance of the investigational IOL to a commercially available monofocal IOL.

ELIGIBILITY:
Key Inclusion Criteria:

* Corrected distance visual acuity (CDVA) worse than 20/40, or presence of visually significant lens opacity;
* Preoperative or predicted postoperative astigmatism of ≤ 1.0 diopter (D);
* Calculated IOL power within range.

Key Exclusion Criteria:

* Current medication that may affect accommodation;
* Systemic disease or concomitant medication that may increase operative risk or confound results;
* Ocular conditions that may predispose the subject for future complications;
* Monocular subjects or subjects with significant permanent visual function loss in fellow eye;
* Previous intraocular or corneal surgery in either eye that may confound the results or increase the risk to the subject, including implantation of a multifocal IOL or other presbyopic corrective surgery in the fellow eye;
* Grade 4 cataract of any type.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Accommodative Amplitude (AA) | Month 6 postoperative
  Accommodative amplitude is the ability of the eye to change its focus from distant to near objects.
Distance Corrected Visual Acuity | Month 6 postoperative
  Visual acuity was measured with distance correction (plus or minus power) in place.
International Organization for Standardization (ISO)-defined Cumulative and Persistent Adverse Events for Posterior Chamber IOL | Up to Month 6 postoperative
  Adverse events were categorized per ISO 11979-7: Ophthalmic Implants - Intraocular Lenses - Part 7: Clinical Investigations.

SECONDARY OUTCOMES:
Accommodative Amplitude | Month 3 postoperative
  Accommodative amplitude is a measure of the range of vision with good acuity.
Minimum Add Power Required to Achieve Best Corrected Near Visual Acuity | Up to Month 6 postoperative
  Plus lenses were placed over the subject's best distance manifest correction.
Uncorrected Visual Acuity | Up to Month 6 postoperative
  Visual acuity was measured without correction in place.

IPD SHARING:
Plan to Share IPD: No